CLINICAL TRIAL: NCT05999435
Title: A DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, ADAPTIVE PHASE 2/3 STUDY OF THE EFFICACY OF LAU-7b IN THE TREATMENT OF ADULTS WITH LONG COVID AND MODERATE TO SEVERE SYMPTOMS
Brief Title: Study of LAU-7b for the Treatment of Long COVID in Adults
Acronym: ESSOR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laurent Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAU-23-01
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
Keywords: Long COVID; COVID-19; Antiviral; Inflammation control
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Fenretinide; Sugars

STUDY DESIGN:
Intervention Model Description: Parallel, regimen-finding, adaptive design well-controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identically appearing active and placebo capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LAU-7b for 3 cycles (Experimental): Each study arm will consist of three (3) cycles of 14 days of treatment intake each spaced by a treatment holiday of 14 days.
  Interventions: Drug: LAU-7b for 3 cycles
- LAU-7b for 1 cycle, then placebo (Experimental): Each study arm will consist of three (3) cycles of 14 days of treatment intake each spaced by a treatment holiday of 14 days.
  Interventions: Drug: LAU-7b for 1 cycle, then placebo
- Placebo for 3 cycles (Placebo Comparator): Each study arm will consist of three (3) cycles of 14 days of treatment intake each spaced by a treatment holiday of 14 days.
  Interventions: Other: Placebo for 3 cycles

INTERVENTIONS:
Drug: LAU-7b for 3 cycles — Three cycles of 14 days of once-a-day intake of LAU-7b, each followed by a treatment intake pause of 14 days.
  Other Names: fenretinide
  Arms: LAU-7b for 3 cycles
Drug: LAU-7b for 1 cycle, then placebo — One cycle of 14 days of once-a-day intake of LAU-7b followed by two cycles of 14 days of placebo administered similarly, each followed by a treatment intake pause of 14 days.
  Other Names: fenretinide
  Arms: LAU-7b for 1 cycle, then placebo
Other: Placebo for 3 cycles — Three cycles of 14 days of once-a-day intake of placebo, each followed by a treatment intake pause of 14 days
  Other Names: sugar pill
  Arms: Placebo for 3 cycles

SUMMARY:
ESSOR is a double-blind, placebo-controlled study of the orally-administered antiviral and inflammation-controlling LAU-7b for the treatment of adults with Long COVID and moderate to severe symptoms.

DETAILED DESCRIPTION:
ESSOR is a multicenter, randomized, double-blind, placebo-controlled Phase 2/3 study of LAU-7b for the treatment of Long COVID in non-hospitalized adults with moderate to severe Long COVID symptoms.

The goal of the study is to evaluate the efficacy of LAU-7b therapy + stable symptomatic standard-of-care relative to placebo + stable symptomatic standard-of-care at reducing the overall Long COVID burden by improving multiple dimensions of quality-of-life and alleviating the symptoms.

This study is a logical extension of investigating LAU-7b as a potential therapeutic against various phases of COVID-19.

LAU-7b is therefore being proposed as a potential disease-modifying medication for the treatment of Long COVID.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years and older, of either gender, and able to give informed consent;
2. Subjects diagnosed with Long COVID and exhibiting persisting, relapsing or new Long COVID symptom(s) at least 12 weeks beyond the start (test positivity or symptom onset) of the causative COVID-19 infection;
3. At least one of the Long COVID symptoms must be from the core list of Long COVID symptoms, and be present for a minimum of 2 weeks prior to screening and of moderate or severe intensity as per the 4-level Likert severity scale (0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms);
4. If female, must be either post-menopausal (one year or greater without menses), surgically sterile, or, for female subjects of child-bearing potential who are capable of conception, must be: practicing a highly effective method of birth control (acceptable methods include intrauterine device, complete abstinence, spermicide + barrier, male partner surgical sterilization, or hormonal contraception) during the study treatment intake and through 30 days after the last dose of the study medication. Periodical abstinence is not classified as an effective method of birth control. A pregnancy test for female subjects of child-bearing potential must be negative at the Screening Visit;
5. Subjects deemed capable of adequate compliance including attending scheduled follow-up calls/visits for the duration of the study, have internet access and able to read and answer questionnaires on electronic Patient Reported Outcomes platform (ePRO) or paper;
6. Screening laboratory test and vital signs results within ranges compatible with the subject's health condition, as per investigator's judgement. See also the last exclusion for certain liver function tests;
7. Subjects deemed capable of swallowing the study treatment capsules

Exclusion Criteria:

1. Subject is currently hospitalized (any reason);
2. Pregnancy or breastfeeding;
3. Any COVID vaccination within 4 weeks of screening or planned during study participation;
4. Presence of any health condition judged by the investigator to be directly causing one or more of the most common Long COVID symptoms;
5. Health condition deemed to possibly interfere with the study endpoints and/or the safety of the subjects. For example, the following conditions should be considered contraindicated for participation in the study. In case of doubt, the Investigator should consult with the Sponsor's medical representative:

   * Febrile neutropenia;
   * Fibromyalgia deemed to interfere with generalized pain measurements;
   * Presence of end-stage cancer (palliative care).
6. Presence or suspicion of drug or alcohol abuse, as judged by the Investigator;
7. Known history of a severe allergy or sensitivity to retinoids, or with known allergies to excipients in the oral capsule formulation proposed to be used in the study;
8. Participation in another interventional drug, alimentary supplement, psychological or device...etc. clinical trial within 30 days (or a minimum of 5 elimination half-lives for drugs) prior to screening, except ongoing participation in non-interventional studies;
9. Presence of total bilirubin >1.5 x Upper Limit of Normal (in the absence of demonstrated Gilbert's syndrome), alanine aminotransferase and/or aspartate aminotransferase > 2.5 x Upper Limit of Normal (unless there are clinical evidences of hepatic steatosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Houle, PhD, Study Director — Laurent Pharmaceuticals Inc.
Locations (5):
- Canada (5):
  - CIUSS du Saguenay-Lac-St-Jean - Hôpital Chicoutimi, Chicoutimi, Quebec
  - Institut de Recherches Cliniques de Montréal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Diex Recherche Québec Inc., Québec, Quebec
  - Centre Hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 specialized Long COVID medical clinics in Quebec. A total of 285 potential participants were screened from 15 November 2023 to 07 May 2024
Groups:
- LAU-7b for 3 Cycles (Arm 1, AAA): Three cycles of 14 days of once-a-day intake of LAU-7b, each followed by a treatment intake pause of 14 days.
- LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP): One cycle of 14 days of once-a-day intake of LAU-7b followed by two cycles of 14 days of placebo administered similarly, each followed by a treatment intake pause of 14 days.
- Placebo for 3 Cycles (Arm 3, PPP): Three cycles of 14 days of once-a-day intake of placebo, each followed by a treatment intake pause of 14 days
Period: Overall Study
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Started (Intent-to-Treat (ITT) population, all participants randomized whether or not receiving the study treatment) | 91 | 91 | 90
Completed | 88 | 90 | 90
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP) | Total
Number analyzed (Participants) | 91 | 91 | 90 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (9.26) | 46.8 (10.96) | 46.5 (10.08) | 47.8 (10.20)
Age, Customized [Count of Participants; unit: Participants]
  Age categories: 18 to 44 years | 24 | 40 | 37 | 101
  Age categories: 45 to 54 years | 39 | 33 | 34 | 106
  Age categories: Equal or greater than 55 years | 28 | 18 | 19 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 78 | 74 | 228
  Male | 15 | 13 | 16 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 91 | 89 | 88 | 268
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 90 | 90 | 89 | 269
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 91 | 91 | 90 | 272
Body Weight [Mean (Standard Deviation); unit: kilograms] | 77.18 (18.972) | 75.98 (17.375) | 81.88 (23.682) | 78.34 (20.264)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter] | 28.14 (7.07) | 27.91 (6.29) | 29.54 (7.82) | 28.53 (7.10)
Vaccinated against Coronavirus Disease 2019 (COVID-19) [Count of Participants; unit: Participants]
  Vaccinated | 87 | 81 | 85 | 253
  Non-vaccinated | 4 | 10 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Physical Component Summary (PCS) of the Medical Outcomes Study Short-Form-36 (SF-36) at Week 12
Description: The SF-36 questionnaire consists of 36 items grouped in eight health domains, vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health, that can be aggregated to two summary scales, physical component summary (PCS ) and mental component summary (MCS). The PCS summarizes the physical status and constitutes the primary outcome variable. Each health domain score consists of the sum scores of the assigned questions. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, ie, severe disability) to 100 (no health restrictions). A higher score means a better physical status. The calculation process for the PCS has been previously described by Taft et al. 2001.
Time Frame: Week 0 and 12
Population: Intent-to-Treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
score on a scale
  PCS at Week 12: number analyzed (Participants) | 88 | 90 | 90
  PCS at Week 12 | 29.47 (9.267) | 29.90 (7.941) | 30.06 (9.484)
  Change from Baseline PCS: number analyzed (Participants) | 85 | 85 | 87
  Change from Baseline PCS | 1.94 (8.034) | 3.32 (7.777) | 2.78 (8.298)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; statistical results of "observed PCS" and "change from baseline PCS are identical; Test type: Superiority; p = 0.4463, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.8, Standard Error of Mean 1.10
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; statistical results of "observed PCS" and "change from baseline PCS are identical; Test type: Superiority; p = 0.8707, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.2, Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Null hypothesis of no difference; statistical results of "observed PCS" and "change from baseline PCS are identical; Test type: Superiority; p = 0.3600, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -1.0, Standard Error of Mean 1.11

2. Secondary Outcome: Safety of LAU-7b, Overview
Description: Number of participants with adverse events. The safety was assessed through the monitoring of adverse events including laboratory test abnormalities, serious adverse events and adverse events leading to study treatment discontinuation. Treatment-emergent adverse event is defined as any adverse event with onset date on or after the first dose of study drug and on or before the Week 12 in person follow-up or until early termination or death, whichever occurred first.
Time Frame: From Week 0 to Week 12
Population: Safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 90 | 91 | 90
participants
  Participants with treatment-emergent adverse events | 71 | 71 | 61
  Participants with serious treatment-emergent adverse events | 1 | 2 | 2
  Participants with treatment-emergent adverse events leading to treatment discontinuation | 7 | 0 | 1
  Participants with treatment-emergent adverse events with fatal outcome | 0 | 0 | 0
  Participants with suspected unexpected serious adverse reaction (SUSAR) | 0 | 0 | 0

3. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: The PGI-C is a single item questionnaire that asks: "Overall, how would you rate the change in your ability to perform usual daily activities since you started the study?".
  These are the 7-point scale options: 1) "very much better", 2) "much better", 3) "minimally better", 4) "no change", 5) "minimally worse", 6) "much worse", or 7) "very much worse".
  Higher scores indicate a change for the worse and lower scores indicate a change for the better.
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  PGI-C at Week 4: number analyzed (Participants) | 87 | 88 | 85
  PGI-C at Week 4: Very much improved | 0 | 1 | 1
  PGI-C at Week 4: Much improved | 10 | 3 | 3
  PGI-C at Week 4: Minimally improved | 25 | 25 | 25
  PGI-C at Week 4: No change | 43 | 46 | 47
  PGI-C at Week 4: Minimally worse | 6 | 7 | 6
  PGI-C at Week 4: Much worse | 2 | 3 | 1
  PGI-C at Week 4: Very much worse | 1 | 3 | 2
  PGI-C at Week 8: number analyzed (Participants) | 87 | 89 | 85
  PGI-C at Week 8: Very much improved | 3 | 0 | 3
  PGI-C at Week 8: Much improved | 11 | 5 | 1
  PGI-C at Week 8: Minimally improved | 23 | 28 | 32
  PGI-C at Week 8: No change | 39 | 42 | 35
  PGI-C at Week 8: Minimally worse | 8 | 8 | 10
  PGI-C at Week 8: Much worse | 2 | 6 | 3
  PGI-C at Week 8: Very much worse | 1 | 0 | 1
  PGI-C at Week 12: number analyzed (Participants) | 88 | 90 | 90
  PGI-C at Week 12: Very much improved | 7 | 0 | 2
  PGI-C at Week 12: Much improved | 9 | 5 | 13
  PGI-C at Week 12: Minimally improved | 18 | 37 | 30
  PGI-C at Week 12: No change | 43 | 38 | 29
  PGI-C at Week 12: Minimally worse | 8 | 5 | 11
  PGI-C at Week 12: Much worse | 2 | 5 | 4
  PGI-C at Week 12: Very much worse | 1 | 0 | 1

4. Secondary Outcome: Proportion of Participants With Marked Improvement in PGI-C
Description: Marked improvement includes "Very much improved" and Much improved". The PGI-C is a single item questionnaire that asks: "Overall, how would you rate the change in your ability to perform usual daily activities since you started the study?".
  These are the 7-point scale options: 1) "very much better", 2) "much better", 3) "minimally better", 4) "no change", 5) "minimally worse", 6) "much worse", or 7) "very much worse".
  Higher scores indicate a change for the worse and lower scores indicate a change for the better.
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Marked improvement of PGI-C at Week 4: number analyzed (Participants) | 87 | 88 | 85
  Marked improvement of PGI-C at Week 4: Participants achieving a marked improvement | 10 | 4 | 4
  Marked improvement of PGI-C at Week 4: No marked improvement | 77 | 84 | 81
  Marked improvement of PGI-C at Week 8: number analyzed (Participants) | 87 | 89 | 85
  Marked improvement of PGI-C at Week 8: Participants achieving a marked improvement | 14 | 5 | 4
  Marked improvement of PGI-C at Week 8: No marked improvement | 73 | 84 | 81
  Marked improvement of PGI-C at Week 12: number analyzed (Participants) | 88 | 90 | 90
  Marked improvement of PGI-C at Week 12: Participants achieving a marked improvement | 16 | 5 | 15
  Marked improvement of PGI-C at Week 12: No marked improvement | 72 | 85 | 75
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1618, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1027, Fisher Exact
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0229, Fisher Exact
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0296, Fisher Exact
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.8448, Fisher Exact
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0307, Fisher Exact
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0105, Fisher Exact

5. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scale
Description: This instrument was developed to characterize fatigue, in cancer and used in other conditions with a phenotype of fatigue. It is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The recall period is 7 days and the response scale employs a 5-point Likert-type scale. The final total score is the sum of the responses for all 13 items and can range from 0 to 52. A higher score means less fatigue.
Time Frame: Weeks 0, 4, 8 and 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
units on a scale
  Value at baseline | 15.68 (8.141) | 15.18 (6.940) | 16.48 (8.456)
  Value at Week 4 | 20.28 (11.524) | 17.77 (9.499) | 19.33 (9.930)
  Change from baseline at Week 4 | 4.70 (8.535) | 2.67 (7.005) | 2.91 (8.103)
  Value at Week 8 | 21.67 (12.426) | 18.20 (9.309) | 19.60 (10.140)
  Change from baseline at Week 8 | 5.94 (8.535) | 3.14 (8.099) | 3.29 (9.057)
  Value at Week 12 | 20.63 (11.914) | 19.07 (9.547) | 22.19 (11.082)
  Change from baseline at Week 12 | 5.07 (8.507) | 4.07 (7.998) | 5.73 (10.749)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2217, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 1.6, Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6834, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.5, Standard Error of Mean 1.30
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1061, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 2.1, Standard Error of Mean 1.31
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0854, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 2.2, Standard Error of Mean 1.30
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6686, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.6, Standard Error of Mean 1.30
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0331, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 2.8, Standard Error of Mean 1.31
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4327, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -1.0, Standard Error of Mean 1.29
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1247, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -2.0, Standard Error of Mean 1.29
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4606, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 1.0, Standard Error of Mean 1.31

6. Secondary Outcome: Change From Baseline in the DePaul Post-Exertional Malaise Questionnaire (DPEMQ)
Description: This instrument was developed to characterize and evaluate the debilitation caused by a physical exertion, whether a usual daily activity or a leisure activity. It is a 10-item questionnaire that assess both the nature of post-exertional malaise (PEM) and duration of symptom. In this study, the presence or not of PEM (based on frequency and severity of 5 PEM items) is determined by the questionnaire. The endpoint of the study is the proportion of participants with PEM at baseline and Week 12, compared between treatment groups.
Time Frame: Weeks 0 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Baseline: number analyzed (Participants) | 88 | 90 | 90
  Baseline: Participants with PEM | 81 | 87 | 84
  Baseline: Participants without PEM | 7 | 3 | 6
  Week 12: number analyzed (Participants) | 87 | 90 | 90
  Week 12: Participants with PEM | 80 | 82 | 83
  Week 12: Participants without PEM | 7 | 8 | 7
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Baseline comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7807, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Baseline comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4965, Fisher Exact — Alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Baseline comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2093, Fisher Exact — Alpha set at 0.05
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05

7. Secondary Outcome: Change From Baseline in Physical Component Summary (PCS) of the Medical Outcomes Study Short-Form-36 (SF-36) at Weeks 4 and 8
Description: The SF-36 questionnaire consists of 36 items grouped in eight health domains, vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health, that can be aggregated to two summary scales, physical component summary (PCS ) and mental component summary (MCS). The PCS summarizes the physical status and constitutes the primary outcome variable. Each health domain score consists of the sum scores of the assigned questions. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, ie, severe disability) to 100 (no health restrictions). A higher score means a better physical status. The calculation process for the PCS has been previously described by Taft et al. 2001. The analysis is performed jointly with the primary outcome measure (Week 12). A positive change from baseline value means improvement, negative value means worsening.
Time Frame: Weeks 0, 4 and 8
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
units on a scale
  PCS at Week 4: number analyzed (Participants) | 87 | 88 | 83
  PCS at Week 4 | 28.71 (6.934) | 29.18 (8.350) | 28.20 (8.767)
  Change from baseline PCS at Week 4: number analyzed (Participants) | 83 | 83 | 82
  Change from baseline PCS at Week 4 | 1.26 (6.950) | 2.89 (7.514) | 1.05 (7.661)
  PCS at Week 8: number analyzed (Participants) | 86 | 89 | 85
  PCS at Week 8 | 30.35 (9.333) | 29.39 (8.295) | 29.64 (9.051)
  Change from baseline PCS at Week 8: number analyzed (Participants) | 83 | 84 | 82
  Change from baseline PCS at Week 8 | 2.64 (8.806) | 2.81 (7.117) | 2.28 (7.897)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7052, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.4, Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1150, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 1.8, Standard Error of Mean 1.11
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2296, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -1.3, Standard Error of Mean 1.11
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7761, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.3, Standard Error of Mean 1.11
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.8544, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.2, Standard Error of Mean 1.11
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.9197, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.1, Standard Error of Mean 1.11

8. Secondary Outcome: Change From Baseline in the Other Aspects (Domain Scales) Than the PCS of the Medical Outcomes Study Short-Form-36 (SF-36)
Description: The SF-36 questionnaire consists of 36 items grouped in eight health domains, vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health, that can be aggregated to two summary scales, physical component summary (PCS ) and mental component summary (MCS). Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, ie, severe disability) to 100 (no health restrictions). A higher score means a better outcome. The study endpoint is the change from baseline in score, a positive change from baseline value means improvement and a negative value means worsening outcome. For sake of conciseness, only Week 12 comparisons are presented.
Time Frame: Weeks 0, 4, 8 and 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
units on a scale
  Baseline vitality score | 17.6 (14.36) | 14.8 (12.55) | 18.8 (14.61)
  Change from baseline vitality score at Week 4 | 7.6 (16.64) | 7.2 (14.61) | 3.9 (15.38)
  Change from baseline vitality score at Week 8 | 10.6 (18.25) | 5.8 (14.74) | 6.2 (18.54)
  Change from baseline vitality score at Week 12 | 7.1 (17.78) | 6.9 (14.23) | 7.8 (19.64)
  Baseline physical functioning score | 42.8 (22.85) | 38.1 (20.55) | 41.6 (23.68)
  Change from baseline physical functioning score at Week 4 | -0.5 (21.19) | 5.8 (21.36) | -1.7 (22.09)
  Change from baseline physical functioning score at Week 8 | 3.9 (24.65) | 4.8 (23.31) | 2.2 (25.05)
  Change from baseline physical functioning score at Week 12 | 3.1 (26.71) | 8.0 (26.95) | 4.6 (25.69)
  Baseline bodily pain score | 35.7 (24.45) | 37.5 (23.44) | 35.3 (22.04)
  Change from baseline bodily pain score at Week 4 | 2.4 (20.50) | 0.4 (21.16) | 3.7 (15.09)
  Change from baseline bodily pain score at Week 8 | 6.2 (19.87) | 3.0 (20.85) | 6.3 (17.94)
  Change from baseline bodily pain score at Week 12 | 4.1 (18.92) | 4.2 (18.35) | 12.0 (24.68)
  Baseline general health perception score | 30.0 (15.80) | 31.4 (14.96) | 31.8 (16.65)
  Change from baseline general health perception score at Week 4 | 3.6 (11.85) | 2.0 (11.20) | 0.8 (12.45)
  Change from baseline general health perception score at Week 8 | 5.1 (13.85) | 1.9 (11.66) | 1.2 (13.05)
  Change from baseline general health perception score at Week 12 | 5.4 (14.57) | 3.4 (13.33) | 2.3 (14.61)
  Baseline physical role functioning score | 1.7 (8.30) | 0.8 (4.54) | 3.7 (14.45)
  Change from baseline physical role functioning score at Week 4 | 3.0 (17.20) | 4.5 (16.99) | 3.0 (23.37)
  Change from baseline physical role functioning score at Week 8 | 7.5 (23.01) | 5.0 (18.82) | 6.4 (26.30)
  Change from baseline physical role functioning score at Week 12 | 2.9 (17.00) | 2.3 (11.90) | 4.3 (20.95)
  Baseline emotional role functioning | 47.0 (45.38) | 55.8 (46.00) | 51.5 (44.61)
  Change from baseline emotional role functioning score at Week 4 | -2.4 (44.41) | -10.3 (45.40) | -5.3 (38.66)
  Change from baseline emotional role functioning score at Week 8 | 6.4 (49.79) | -6.7 (46.80) | -0.4 (44.90)
  Change from baseline emotional role functioning score at Week 12 | 1.6 (48.50) | -6.6 (43.93) | 6.9 (43.37)
  Baseline social role functioning score | 23.9 (19.66) | 23.3 (19.06) | 26.6 (19.68)
  Change from baseline social role functioning score at Week 4 | 5.6 (18.95) | 3.9 (17.56) | 4.4 (16.82)
  Change from baseline social role functioning score at Week 8 | 10.4 (20.08) | 5.4 (18.94) | 7.2 (19.15)
  Change from baseline social role functioning score at Week 12 | 10.4 (21.12) | 7.6 (20.15) | 9.3 (23.75)
  Baseline mental health score | 55.7 (6.28) | 56.1 (8.11) | 56.2 (8.05)
  Change from baseline mental health score at Week 4 | 1.0 (7.04) | -0.2 (7.62) | 1.3 (7.98)
  Change from baseline mental health score at Week 8 | 0.7 (6.89) | -0.2 (7.40) | 0.7 (7.09)
  Change from baseline mental health score at Week 12 | 1.0 (7.66) | -0.0 (8.45) | -0.1 (7.92)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Vitality domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6269, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -1.2, Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Vitality domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4427, Mixed Models Analysis — Alpha set at 0.05; Leat Square Means difference = -1.9, Standard Error of Mean 2.50
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Vitality domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7783, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 0.7, Standard Error of Mean 2.52
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7488, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -1.0, Standard Error of Mean 3.19
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.5557, Mixed Models Analysis; Least Square Means difference = 1.9, Standard Error of Mean 3.18
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3679, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -2.9, Standard Error of Mean 3.22
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Bodily Pain domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0044, Mixed Models Analysis — Alpha set at 0.05; Least Squre Means difference = -8.0, Standard Error of Mean 2.78
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Bodily Pain domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0158, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -6.8, Standard Error of Mean 2.79
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Bodily Pain domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6682, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -1.2, Standard Error of Mean 2.81
Statistical Analysis 10: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); General Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2448, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 2.2, Standard Error of Mean 1.90
Statistical Analysis 11: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); General Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4702, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 1.4, Standard Error of Mean 1.90
Statistical Analysis 12: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); General Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6627, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 0.8, Standard Error of Mean 1.92
Statistical Analysis 13: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Role Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2774, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -3.1, Standard Error of Mean 2.85
Statistical Analysis 14: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Role Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1537, Mixed Models Analysis; Least Square Means difference = -4.1, Standard Error of Mean 2.85
Statistical Analysis 15: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Role Physical Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7355, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 1.0, Standard Error of Mean 2.87
Statistical Analysis 16: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Role Emotional Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1757, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -8.0, Standard Error of Mean 5.90
Statistical Analysis 17: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Rome Emotional Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0649, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -10.9, Standard Error of Mean 5.89
Statistical Analysis 18: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Role Emotional Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6262, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 2.9, Standard Error of Mean 5.93
Statistical Analysis 19: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Social Role Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.9709, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 0.1, Standard Error of Mean 2.92
Statistical Analysis 20: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Social Role Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3201, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -2.9, Standard Error of Mean 2.92
Statistical Analysis 21: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Social Role Functioning domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3065, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 3.0, Standard Error of Mean 2.95
Statistical Analysis 22: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Mental Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2891, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 1.0, Standard Error of Mean 0.95
Statistical Analysis 23: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Mental Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.8714, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = -0.2, Standard Error of Mean 0.95
Statistical Analysis 24: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Mental Health domain, Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2260, Mixed Models Analysis — Alpha set at 0.05; Least Square Means difference = 1.2, Standard Error of Mean 0.96

9. Secondary Outcome: Proportion of Subjects Who Judge to Have Regained Their Daily Usual Activity Level of Pre-causative-infection.
Description: This will be assessed by a single question with either yes or no as answer: "Do you judge that you have regained the daily usual activity level you had prior to being infected by COVID-19 back in Month xxxx? By daily usual activity we mean work, leisure, physical exercise...etc."
Time Frame: From Week 0 through Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Week 4: number analyzed (Participants) | 89 | 91 | 90
  Week 4: Participants who judge to have regained daily usual activity level | 0 | 3 | 0
  Week 4: Participants who judge NOT to have regained daily usual activity level | 89 | 88 | 90
  Week 8: number analyzed (Participants) | 88 | 90 | 90
  Week 8: Participants who judge to have regained daily usual activity level | 0 | 0 | 1
  Week 8: Participants who judge NOT to have regained daily usual activity level | 88 | 90 | 89
  Week 12: number analyzed (Participants) | 88 | 90 | 90
  Week 12: Participants who judge to have regained daily usual activity level | 0 | 1 | 2
  Week 12: Participants who judge NOT to have regained daily usual activity level | 88 | 89 | 88
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; No comparison possible since zero count in both groups
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2459, Fisher Exact — Alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2459, Fisher Exact — Alpha set at 0.05
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; No comparison possible since zero count in both groups
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4972, Fisher Exact — Alpha set to 0.05
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact

10. Secondary Outcome: Proportion of Subjects Achieving >=25% (>=50% and >=75% Presented Separately) Improvement in the Sum of Individual Core Long COVID Symptom Severity as Evaluated by a Standard 4-level Likert Scale.
Description: The Core (most common) Long COVID symptoms are: fatigue, trouble sleeping, shortness of breath, general pain and discomfort, cognitive problems (most commonly known as brain fog or memory fog) and mental health symptoms.
  Each symptom is rated as: 0=No symptom, 1=Mild symptom (no interference with daily activities), 2=Moderate symptom (interfere and may limit daily activities), and 3=Severe symptom (strong interference preventing daily activities. The higher the rating is, worse is the symptom.
  0 and 1 are deemed not burdensome, 2 and 3 are burdensome. A sum of the burdensome category is calculated for each visit and is the endpoint being evaluated for improvement since burdensome symptoms are those with highest impact on daily usual activity level.
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Week 4: number analyzed (Participants) | 89 | 90 | 90
  Week 4: Participants with at least 25% improvement in burdensome symptoms total score | 10 | 6 | 6
  Week 4: Participants not reaching 25% improvement in burdensome symptoms total score | 79 | 84 | 84
  Week 8: number analyzed (Participants) | 83 | 90 | 88
  Week 8: Participants with at least 25% improvement in burdensome symptoms total score | 15 | 18 | 7
  Week 8: Participants not reaching 25% improvement in burdensome symptoms total score | 68 | 72 | 81
  Week 12: number analyzed (Participants) | 85 | 89 | 88
  Week 12: Participants with at least 25% improvement in burdensome symptoms total score | 15 | 16 | 18
  Week 12: Participants not reaching 25% improvement in burdensome symptoms total score | 70 | 73 | 70
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3081, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3081, Fisher Exact
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.066, Fisher Exact — Alpha set at 0.05
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0297, Fisher Exact — Alpha set at 0.05
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.8471, Fisher Exact — Alpha set at 0.05
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7009, Fisher Exact — Alpha set at 0.05
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7064, Fisher Exact — Alpha set at 0.05
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05

11. Secondary Outcome: Proportion of Subjects Achieving >=50% (>=25% and >=75% Presented Separately) Improvement in the Sum of Individual Core Long COVID Symptom Severity as Evaluated by a Standard 4-level Likert Scale.
Description: as for outcome 10
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Week 4: number analyzed (Participants) | 89 | 90 | 90
  Week 4: Participants with at least 50% improvement in burdensome symptoms total score | 6 | 1 | 2
  Week 4: Participants not reaching 50% improvement in burdensome symptoms total score | 83 | 89 | 88
  Week 8: number analyzed (Participants) | 83 | 90 | 88
  Week 8: Participants with at least 50% improvement in burdensome symptoms total score | 9 | 3 | 4
  Week 8: Participants not reaching 50% improvement in burdensome symptoms total score | 74 | 87 | 84
  Week 12: number analyzed (Participants) | 85 | 89 | 88
  Week 12: Participants with at least 50% improvement in burdensome symptoms total score | 7 | 3 | 10
  Week 12: Participants not reaching 50% improvement in burdensome symptoms total score | 78 | 86 | 78
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1686, Fisher Exact
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0643, Fisher Exact — Alpha set at 0.05
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1531, Fisher Exact
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7187, Fisher Exact
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0720, Fisher Exact — Alpha set at 0.05
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6117, Fisher Exact — Alpha set at 0.05
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0479, Fisher Exact — Alpha set at 0.05
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2042, Fisher Exact — Alpha set at 0.05

12. Secondary Outcome: Proportion of Subjects Achieving >=75% (>=25% and >=50% Presented Separately) Improvement in the Sum of Individual Core Long COVID Symptom Severity as Evaluated by a Standard 4-level Likert Scale.
Description: as for outcome 10
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Week 4: number analyzed (Participants) | 89 | 90 | 90
  Week 4: Participants with at least 75% improvement in burdensome symptoms total score | 2 | 0 | 0
  Week 4: Participants not reaching 75% improvement in burdensome symptoms total score | 87 | 90 | 90
  Week 8: number analyzed (Participants) | 83 | 90 | 88
  Week 8: Participants with at least 75% improvement in burdensome symptoms total score | 1 | 0 | 1
  Week 8: Participants not reaching 75% improvement in burdensome symptoms total score | 82 | 90 | 87
  Week 12: number analyzed (Participants) | 85 | 89 | 88
  Week 12: Participants with at least 75% improvement in burdensome symptoms total score | 1 | 0 | 1
  Week 12: Participants not reaching 75% improvement in burdensome symptoms total score | 84 | 89 | 87
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2458, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; Comparison not possible since zero counts in both groups
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.2458, Fisher Exact
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4944, Fisher Exact — Alpha set at 0.05
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4798, Fisher Exact
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4972, Fisher Exact — Alpha set at 0.05
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4885, Fisher Exact — Alpha set at 0.05

13. Secondary Outcome: Change From Baseline in the EuroQol-5 Dimensions -5 Levels (EQ-5D-5L) Score
Description: EQ-5D-5L is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). Higher values indicate worse outcomes, while lower indicate better outcomes. The subscales are combined to compute a total score index, adjusted for a standard value of general population in a country/region and averaged to produce the mean and SD. The Summary index value range is from 0 to 1, where 1 is considered the best possible health and 0 is the worst possible health. For the change in score, a positive number indicates that the scores improved from baseline.
Time Frame: Weeks 0, 4, 8 and 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
score on a scale
  Baseline Summary Index | 0.60 (0.195) | 0.56 (0.209) | 0.58 (0.213)
  Change from baseline at Week 4 | 0.01 (0.178) | 0.03 (0.164) | 0.04 (0.150)
  Change from baseline at Week 8 | 0.03 (0.158) | 0.02 (0.188) | 0.03 (0.174)
  Change from baseline at Week 12 | 0.04 (0.150) | 0.03 (0.168) | 0.08 (0.187)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4156, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7088, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6610, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7580, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.0, Standard Error of Mean 0.02
Statistical Analysis 5: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.4974, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 6: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.3289, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.0, Standard Error of Mean 0.02
Statistical Analysis 7: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.1700, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 8: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.0557, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = -0.0, Standard Error of Mean 0.02
Statistical Analysis 9: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6008, Mixed Models Analysis — No adjustment for multiple comparisons, alpha set at 0.05; Least Square Means difference = 0.0, Standard Error of Mean 0.02

14. Secondary Outcome: Proportion of Subjects With Relief of at Least One Core Burdensome Long COVID Symptom for a Minimum of 2 Weeks.
Description: The core Long COVID symptoms are: fatigue, trouble sleeping, shortness of breath, general pain and discomfort, cognitive problems (most commonly known as brain fog or memory fog) and mental health symptoms.
  Each symptom is rated as: 0=No symptom, 1=Mild symptom (no interference with daily activities), 2=Moderate symptom (interfere and may limit daily activities), and 3=Severe symptom (strong interference preventing daily activities. The higher the rating is, worse is the symptom.
  0 and 1 are deemed not burdensome, 2 and 3 are burdensome.
  Relief means a reduction of severity from moderate to none, or severe to mild/none (≥2-point Likert score change)
Time Frame: From Week 0 to Week 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Participants with relief of at least one core burdensome symptom | 8 | 9 | 9
  Participants without relief of core burdensome symptoms | 83 | 82 | 81
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; Test type: Superiority; p = 0.8046, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05

15. Secondary Outcome: Time to Relief of the First Core Burdensome Long COVID Symptom for a Minimum of 2 Weeks, Among Those Symptoms Present at Baseline.
Description: The core Long COVID symptoms are: fatigue, trouble sleeping, shortness of breath, general pain and discomfort, cognitive problems (brain fog or memory fog) and mental health symptoms. Each symptom is rated as: 0=No symptom, 1=Mild symptom (no interference with daily activities), 2=Moderate symptom (interfere and may limit daily activities), and 3=Severe symptom (strong interference preventing daily activities. The higher the rating is, worse is the symptom. 0 and 1 are deemed not burdensome, 2 and 3 are burdensome. This will be assessed through periodic inventory of the core Long COVID symptoms, performed at each visit. Relief means a reduction of severity from moderate to none, or severe to mild/none (≥2-point Likert score change). A longer time is worse than a short time to resolution.
Time Frame: From Week 0 to Week 12
Population: ITT population, Incidence rate of relief of at least one core burdensome symptom is less than 10%. Kaplan-Meier analysis and estimates, as well as log-rank test are not reliable and were not performed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
days | 60.13 (19.23) | 64.78 (19.38) | 71.67 (14.64)

16. Secondary Outcome: Proportion of Subjects With a Sustained Clinical Recovery, Meaning a Relief of All Core Long COVID Symptoms.
Description: The core Long COVID symptoms are: fatigue, trouble sleeping, shortness of breath, general pain and discomfort, cognitive problems (most commonly known as brain fog or memory fog) and mental health symptoms.
  Each symptom is rated as: 0=No symptom, 1=Mild symptom (no interference with daily activities), 2=Moderate symptom (interfere and may limit daily activities), and 3=Severe symptom (strong interference preventing daily activities. The higher the rating is, worse is the symptom.
  0 and 1 are deemed not burdensome, 2 and 3 are burdensome.
  This will be assessed through periodic inventory of the core Long COVID symptoms, performed at each visit. Relief means a reduction of severity from moderate to none, or severe to mild/none (≥2-point Likert score change). A higher proportion is better than a lower proportion.
Time Frame: Weeks 4, 8 and 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Week 4: number analyzed (Participants) | 89 | 91 | 90
  Week 4: Participants achieving sustained recovery of all core symptoms | 0 | 0 | 0
  Week 4: Participants NOT achieving sustained recovery of all core symptoms | 89 | 91 | 90
  Week 8: number analyzed (Participants) | 88 | 90 | 90
  Week 8: Participants achieving sustained recovery of all core symptoms | 0 | 0 | 0
  Week 8: Participants NOT achieving sustained recovery of all core symptoms | 88 | 90 | 90
  Week 12: number analyzed (Participants) | 88 | 90 | 90
  Week 12: Participants achieving sustained recovery of all core symptoms | 0 | 0 | 0
  Week 12: Participants NOT achieving sustained recovery of all core symptoms | 88 | 90 | 90
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; Test type: Superiority; Sustained recovery was not achieved in any participant, no possible statistical analysis

17. Secondary Outcome: Change From Baseline in the Total Number of Long COVID Symptoms (Core and Non-core).
Description: This will be assessed through periodic inventory of all the Long COVID symptoms, performed at each visit, relative to the baseline inventory. A lower total number is better than a higher total number.
Time Frame: Weeks 0, 4, 8 and 12, as well as the longer term visit at Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: count of symptoms
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
count of symptoms
  Baseline count of all Long COVID symptoms | 14.3 (7.07) | 15.2 (7.98) | 15.0 (7.88)
  Count of all Long COVID symptoms at Week 4: number analyzed (Participants) | 89 | 91 | 90
  Count of all Long COVID symptoms at Week 4 | 14.2 (7.06) | 15.1 (8.04) | 15.0 (7.90)
  Count of all Long COVID symptoms at Week 8: number analyzed (Participants) | 88 | 90 | 90
  Count of all Long COVID symptoms at Week 8 | 14.4 (7.25) | 15.0 (8.07) | 14.9 (7.57)
  Count of all Long COVID symptoms at Week 12: number analyzed (Participants) | 88 | 90 | 90
  Count of all Long COVID symptoms at Week 12 | 14.4 (7.18) | 15.0 (8.05) | 14.9 (7.55)
  Count of all Long COVID symptoms at Week 24: number analyzed (Participants) | 87 | 89 | 90
  Count of all Long COVID symptoms at Week 24 | 14.4 (7.26) | 14.8 (8.20) | 14.7 (7.65)
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 4 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.7699, ANOVA — Treatment group effect, alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 8 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.9928, ANOVA — Treatment group effect, alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 12 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.8363, ANOVA — Treatment group effect, alpha set at 0.05
Statistical Analysis 4: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Week 24 comparison, null hypothesis of no difference; Test type: Superiority; p = 0.6930, ANOVA — Treatment group effect, alpha set at 0.05

18. Secondary Outcome: Proportion of Subjects With Long COVID-related Unplanned Medical Visits
Description: This will be assessed by probing the subjects at each visit. Long COVID-related unplanned medical visits includes visits to practitioner's office, urgent care visits, emergency room <24h, or hospitalization >24 hours.
  A higher proportion is worse than a lower proportion
Time Frame: From Week 0 to Week 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Participants with Long COVID-related unplanned medical visits | 2 | 3 | 5
  Participants without Long COVID-related unplanned medical visits | 89 | 88 | 85
Statistical Analysis 1: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; Test type: Superiority; p = 0.2780, Fisher Exact — Alpha set at 0.05
Statistical Analysis 2: Comparison: LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) vs Placebo for 3 Cycles (Arm 3, PPP); Null hypothesis of no difference; Test type: Superiority; p = 0.4967, Fisher Exact — Alpha set at 0.05
Statistical Analysis 3: Comparison: LAU-7b for 3 Cycles (Arm 1, AAA) vs LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP); Null hypothesis of no difference; Test type: Superiority; p = 1.000, Fisher Exact — Alpha set at 0.05

19. Secondary Outcome: Proportion of Subjects Deceased From Any Cause Through Week 12.
Description: This will be assessed by probing the subjects at each visit, including caretakers or relatives if the subjects cannot be reached at a given visit.
  A higher proportion is worse than a lower proportion
Time Frame: From Week 0 to Week 12
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Participants deceased from any cause through Week 12 | 0 | 0 | 0
  Participants alive through Week 12 | 91 | 91 | 90

20. Secondary Outcome: Proportion of Subjects With Significant Cardiovascular Events
Description: A significant cardiovascular event is one that results in at least an acute care visit, a hospitalization or an event-related death.
  A higher proportion is worse than a lower proportion
Time Frame: From Week 0 to Week 12 and including up to the long-term follow-up at Week 24
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Participants with significant cardiovascular event through Week 24 | 0 | 0 | 0
  Participants without significant cardiovascular event through Week 24 | 91 | 91 | 90

21. Other Pre Specified Outcome: Health and Survival Follow-up (Week 24), Long COVID Symptom Count
Description: This is now presented as part of Outcome #17. Initially planned to be separate from the reporting and analysis of the Week 12 outcomes, a longer term contact was made at Week 24 to assess the following: Presence or not of Long COVID symptoms (total number of Long COVID symptoms).
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: counts of symptoms
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 87 | 89 | 90
counts of symptoms | 14.4 (7.26) | 14.8 (8.20) | 14.7 (7.65)

22. Other Pre Specified Outcome: Health and Survival Follow-up (Week 24), Significant Cardiovascular Events
Description: General health check-up: Assess significant cardiovascular events (one that results in at least an acute care visit, a hospitalization or an event-related death) and survival.
Time Frame: Week 24
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 91 | 91 | 90
Participants
  Participants with significant cardiovascular events or death through Week 24 | 0 | 0 | 0
  Participants without significant cardiovascular events or death through Week 24 | 91 | 91 | 90

23. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Hematologic Function (Except Hemoglobin & Hematocrit)
Description: These will be assessed by blood samples taken at randomization visit in a subgroup of participants consented to contribute samples.
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
cells*10^9/L
  Erythrocyte count (10^9/L) - Baseline | 4496 (442.2) | 4703 (384.7) | 4610 (431.8)
  Leucocyte count (10^9/L) - Baseline | 6.53 (2.102) | 5.99 (1.576) | 6.28 (1.634)
  Platelet count (10^9/L) - Baseline | 265 (75.9) | 261 (56.8) | 252 (73.1)
  Neutrophil count (10^9/L) - Baseline | 4.23 (1.655) | 3.59 (1.307) | 3.95 (1.369)

24. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Hematologic Function (Hemoglobin)
Description: as for outcome 23
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 27 | 25 | 24
g/L | 137 (11.8) | 141 (8.8) | 142 (13.7)

25. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Hematologic Function (Hematocrit)
Description: as for outcome 23
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 27 | 25 | 24
L/L | 0.409 (0.0358) | 0.417 (0.0269) | 0.418 (0.0405)

26. Other Pre Specified Outcome: Changes Relative to Baseline (Percent Change) of Systemic Biomarkers of Hematologic Function
Description: These will be assessed by blood samples taken at specific visits of the study in a subgroup of participants consented to contribute samples.
Time Frame: Weeks 0, 2 and 10
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
Percentage of change
  Erythrocyte % change from baseline at Week 2: number analyzed (Participants) | 25 | 25 | 24
  Erythrocyte % change from baseline at Week 2 | -1.29 (3.267) | -0.98 (4.386) | 0.34 (3.482)
  Erythrocyte % change from baseline at Week 10: number analyzed (Participants) | 22 | 23 | 21
  Erythrocyte % change from baseline at Week 10 | -0.55 (7.443) | -0.44 (4.418) | -1.40 (4.534)
  Leucocyte % change from baseline at Week 2: number analyzed (Participants) | 25 | 25 | 24
  Leucocyte % change from baseline at Week 2 | -2.89 (18.551) | 4.90 (21.194) | 0.05 (19.758)
  Leucocyte % change from baseline at Week 10: number analyzed (Participants) | 22 | 23 | 21
  Leucocyte % change from baseline at Week 10 | 5.70 (37.957) | 5.31 (14.887) | -2.97 (15.053)
  Platelet % change from baseline at Week 2: number analyzed (Participants) | 25 | 25 | 24
  Platelet % change from baseline at Week 2 | -2.90 (10.746) | -3.39 (15.811) | 2.66 (9.501)
  Platelet % change from baseline at Week 10: number analyzed (Participants) | 22 | 23 | 21
  Platelet % change from baseline at Week 10 | -3.14 (12.807) | -2.25 (12.003) | 0.45 (12.018)
  Hematocrit % change at Week 2: number analyzed (Participants) | 25 | 24 | 24
  Hematocrit % change at Week 2 | -1.66 (4.349) | -1.18 (3.988) | 0.26 (3.960)
  Hematocrit % change at Week 10: number analyzed (Participants) | 22 | 22 | 21
  Hematocrit % change at Week 10 | -1.08 (3.956) | -0.41 (4.632) | -1.28 (5.252)
  Hemoglobin % change at Week 2: number analyzed (Participants) | 25 | 25 | 24
  Hemoglobin % change at Week 2 | -1.37 (3.329) | -0.83 (3.194) | -0.51 (3.439)
  Hemoglobin % change at Week 10: number analyzed (Participants) | 22 | 23 | 21
  Hemoglobin % change at Week 10 | -0.74 (4.194) | -0.71 (3.712) | -1.70 (3.910)
  Neutrophil % change at Week 2: number analyzed (Participants) | 25 | 25 | 24
  Neutrophil % change at Week 2 | -6.02 (24.371) | 10.47 (34,679) | -0.22 (27.398)
  Neutrophil % change at Week 10: number analyzed (Participants) | 22 | 23 | 21
  Neutrophil % change at Week 10 | 5.62 (52.222) | 6.71 (25.699) | -6.75 (22.195)

27. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Inflammation and Immunologic Function (Parameters in pg/mL)
Description: These will be assessed by blood samples taken at randomization visits of the study in a subgroup of participants consented to contribute samples.
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
pg/mL
  Baseline Interleukin-1-beta (pg/mL) | 0.347 (0.4324) | 0.439 (0.6867) | 0.197 (0.1472)
  Baseline Interleukin-6 (pg/mL) | 1.880 (1.5469) | 1.316 (0.7612) | 1.424 (0.8999)
  Baseline Interleukin-8 (pg/mL) | 7.984 (5.4974) | 7.174 (4.1427) | 7.619 (4.1476)
  Baseline Interleukin-10 (pg/mL) | 0.470 (0.5790) | 0.308 (0.1848) | 0.282 (0.1825)
  Baseline Interferon-lambda-1 (pg/mL) | 4.800 (5.0653) | 2.886 (1.9873) | 3.837 (2.7632)
  Baseline Interferon-lambda-3 (pg/mL) | 43.006 (15.0238) | 15.015 (2.6113) | 16.589 (0.3848)
  Baseline Interferon-gamma (pg/mL) | 25.235 (68.9460) | 10.449 (12.3146) | 10772 (10.4890)
  Baseline Tumor Necrosis Factor alpha (pg/mL) | 1.593 (1.4729) | 1.093 (0.6115) | 1.210 (0.8951)
  Baseline Cluster of Differentiation 40 ligand (pg/mL) | 1554.382 (1450.9193) | 1570.212 (872.6533) | 2201.813 (1421.8699)
  Baseline Interferon gamma-induced protein 10 (pg/mL) | 394.642 (510.0155) | 331.127 (247.5556) | 257.239 (160.3321)

28. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Inflammation and Immunologic Function (Calprotectin, C-reactive Protein)
Description: as for outcome 27
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
µg/mL
  Baseline Calprotectin (µg/mL) | 1.335 (2.1836) | 1.091 (1.8067) | 1.282 (2.1241)
  Baseline C-reactive protein (µg/mL) | 6.253 (5.9201) | 3.061 (2.6015) | 4.391 (8.5794)

29. Other Pre Specified Outcome: Baseline Values of Systemic Biomarkers of Inflammation and Immunologic Function (Serotonin, Tryptophan and Taurine)
Description: as for outcome 27
Time Frame: Week 0
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
µmol/L
  Baseline Serotonin (µmol/L) | 1.894 (2.3104) | 1.382 (2.4128) | 1.915 (1.9254)
  Baseline Tryptophan (µmol/L) | 56.688 (11.3971) | 58.115 (11.3080) | 55.397 (8.5476)
  Baseline Taurine (µmol/L) | 97.381 (30.2629) | 104.615 (32.5454) | 108.351 (39.1587)

30. Other Pre Specified Outcome: Changes Relative to Baseline (Percent Change) of Systemic Biomarkers of Inflammation and Immunologic Function
Description: as for outcome 26
Time Frame: Weeks 0, 2 and 10
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
Percentage of change
  Interleukin-1-beta % change from baseline at Week 2: number analyzed (Participants) | 21 | 17 | 19
  Interleukin-1-beta % change from baseline at Week 2 | 71.6 (245.5) | 45.9 (207.0) | 19.3 (55.3)
  Interleukin-1-beta % change from baseline at Week 10: number analyzed (Participants) | 18 | 18 | 16
  Interleukin-1-beta % change from baseline at Week 10 | 32.1 (151.1) | -23.6 (32.3) | 176.5 (678.5)
  Interleukin-6 % change from baseline at Week 2: number analyzed (Participants) | 27 | 24 | 24
  Interleukin-6 % change from baseline at Week 2 | 33.6 (138.1) | 30.7 (77.3) | 19.6 (50.6)
  Interleukin-6 % change from baseline at Week 10: number analyzed (Participants) | 23 | 23 | 21
  Interleukin-6 % change from baseline at Week 10 | 38.3 (182.9) | -10.6 (30.8) | 35.7 (165.6)
  Interleukin-8 % change from baseline at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Interleukin-8 % change from baseline at Week 2 | 14.9 (48.3) | 12.9 (29.1) | 27.2 (127.7)
  Interleukin-8 % change from baseline at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Interleukin-8 % change from baseline at Week 10 | 35.6 (59.4) | 19.8 (58.6) | 15.6 (51.3)
  Interleukin-10 % change at Week 2: number analyzed (Participants) | 26 | 25 | 24
  Interleukin-10 % change at Week 2 | 43.6 (119.8) | 43.4 (121.9) | 8.2 (31.0)
  Interleukin-10 % change at Week 10: number analyzed (Participants) | 22 | 24 | 21
  Interleukin-10 % change at Week 10 | 39.3 (125.1) | -14.2 (37.6) | 52.6 (283.2)
  Interferon-lambda-1 % change at Week 2: number analyzed (Participants) | 25 | 25 | 23
  Interferon-lambda-1 % change at Week 2 | 1.1 (46.2) | 19.4 (77.6) | 8.3 (51.0)
  Interferon-lambda-1 % change at Week 10: number analyzed (Participants) | 21 | 23 | 20
  Interferon-lambda-1 % change at Week 10 | 127.0 (152.0) | 90.9 (113.6) | 92.7 (245.1)
  Interferon-lambda-3 % change at Week 2: number analyzed (Participants) | 2 | 2 | 1
  Interferon-lambda-3 % change at Week 2 | -10.5 (10.8) | 10.4 (46.0) | -4.15 (NA) — single observation
  Interferon-lambda-3 % change at Week 10: number analyzed (Participants) | 1 | 2 | 0
  Interferon-lambda-3 % change at Week 10 | -16.9 (NA) — single observation | 87.1 (10.9) |
  Interferon-gamma % change at Week 2: number analyzed (Participants) | 26 | 25 | 22
  Interferon-gamma % change at Week 2 | 43.7 (146.8) | 134.3 (320.8) | 115.4 (513.3)
  Interferon-gamma % change at Week 10: number analyzed (Participants) | 22 | 24 | 19
  Interferon-gamma % change at Week 10 | -16.1 (50.0) | -32.8 (40.8) | 5.4 (86.8)
  Tumor Necrosis Factor alpha % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Tumor Necrosis Factor alpha % change at Week 2 | 112.3 (459.7) | 65.1 (147.5) | 17.0 (59.7)
  Tumor Necrosis Factor alpha % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Tumor Necrosis Factor alpha % change at Week 10 | 76.3 (206.1) | 21.9 (72.2) | 84.9 (187.2)
  Cluster of Differentiation 40 ligand % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Cluster of Differentiation 40 ligand % change at Week 2 | 43.6 (106.3) | 35.7 (106.1) | 60.3 (188.2)
  Cluster of Differentiation 40 ligand % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Cluster of Differentiation 40 ligand % change at Week 10 | 36.1 (100.0) | 36.7 (113.1) | 43.2 (108.8)
  Interferon gamma-induced protein 10 % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Interferon gamma-induced protein 10 % change at Week 2 | 18.0 (68.6) | 37.0 (64.1) | 15.9 (45.6)
  Interferon gamma-induced protein 10 % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Interferon gamma-induced protein 10 % change at Week 10 | -29.5 (35.1) | -32.0 (32.7) | -10.5 (54.3)
  Calprotectin % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Calprotectin % change at Week 2 | 187.7 (658.7) | 159.8 (572.9) | 65.3 (256.0)
  Calprotectin % change at Week 10: number analyzed (Participants) | 23 | 23 | 21
  Calprotectin % change at Week 10 | 9.6 (78.6) | 193.2 (629.7) | 219.1 (615.5)
  C-reactive protein % change at Week 2: number analyzed (Participants) | 13 | 9 | 11
  C-reactive protein % change at Week 2 | 25.2 (95.4) | 185.6 (549.4) | 3.5 (25.7)
  C-reactive protein % change at Week 10: number analyzed (Participants) | 11 | 8 | 9
  C-reactive protein % change at Week 10 | -8.9 (46.1) | 19.3 (55.2) | 71.6 (236.3)
  Serotonin % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Serotonin % change at Week 2 | 10.5 (50.7) | 274.5 (1257.3) | 606.1 (2059.9)
  Serotonin % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Serotonin % change at Week 10 | 51.2 (98.9) | 9.0 (65.3) | 5.1 (96.2)
  Tryptophan % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Tryptophan % change at Week 2 | -1.2 (24.8) | 2.4 (15.3) | 4.4 (21.4)
  Tryptophan % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Tryptophan % change at Week 10 | 8.1 (31.1) | 2.7 (16.0) | 1.2 (18.5)
  Taurine % change at Week 2: number analyzed (Participants) | 27 | 25 | 24
  Taurine % change at Week 2 | 13.1 (38.5) | 13.0 (47.1) | 29.7 (77.0)
  Taurine % change at Week 10: number analyzed (Participants) | 23 | 24 | 21
  Taurine % change at Week 10 | 12.4 (36.2) | 5.6 (38.9) | 18.0 (50.7)

31. Other Pre Specified Outcome: Biomarkers of Pharmacodynamic Activity - Plasma Retinol
Description: as for outcome 26
Time Frame: Weeks 0, 2 and 10
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
µmol/L
  Baseline Retinol (µmol/L): number analyzed (Participants) | 9 | 7 | 4
  Baseline Retinol (µmol/L) | 1.89 (0.389) | 1.92 (0.303) | 2.05 (0.298)
  Week 2 Retinol (µmol/L): number analyzed (Participants) | 8 | 8 | 5
  Week 2 Retinol (µmol/L) | 0.42 (0.198) | 0.39 (0.092) | 1.81 (0.336)
  Week 10 Retinol (µmol/L): number analyzed (Participants) | 9 | 8 | 5
  Week 10 Retinol (µmol/L) | 0.37 (0.097) | 2.08 (0.541) | 2.07 (0.540)

32. Other Pre Specified Outcome: Biomarkers of Pharmacodynamic Activity - Systematic Inflammation Index (SII)
Description: These will be assessed by blood samples taken at specific visits of the study in a subgroup of participants consented to contribute samples. SII = (N × P)/L, where N, P and L (cells*10^9/L) represent absolute neutrophil counts, platelet counts and lymphocyte counts. Since SII is a ratio of concentrations, it is unitless.
Time Frame: Weeks 0, 2 and 10
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: unitless value
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
unitless value
  Baseline Systematic Inflammation Index: number analyzed (Participants) | 27 | 25 | 24
  Baseline Systematic Inflammation Index | 726.4 (358.63) | 545.2 (190.27) | 628.8 (322.79)
  Week 2 Systematic Inflammation Index: number analyzed (Participants) | 25 | 25 | 24
  Week 2 Systematic Inflammation Index | 626.5 (370.06) | 558.9 (169.71) | 632.2 (338.37)
  Week 10 Systematic Inflammation Index: number analyzed (Participants) | 22 | 23 | 21
  Week 10 Systematic Inflammation Index | 639.5 (414.09) | 513.2 (159.02) | 563.5 (336.95)

33. Other Pre Specified Outcome: Changes Relative to Baseline (Percent Change) of Biomarker of Pharmacodynamic Activity - Retinol
Description: as for outcome 26
Time Frame: Weeks 0, 2 and 10
Population: Biomarker subset of participants
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
Number analyzed (Participants) | 28 | 25 | 24
percentage of baseline
  Retinol % change from baseline at Week 2: number analyzed (Participants) | 7 | 7 | 4
  Retinol % change from baseline at Week 2 | -78.9 (5.94) | -79.5 (6.36) | -4.4 (8.24)
  Retinol % change from baseline at Week 10: number analyzed (Participants) | 8 | 7 | 4
  Retinol % change from baseline at Week 10 | -80.8 (4.274) | 0.3 (12.19) | 6.2 (21.15)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the Week 12 in person follow-up, or until early termination or death, whichever occurred first. Treatment emergent adverse events (TEAE) occurred from the first dose of study treatment (or worsened after first dose of study treatment) until the end of the AE collection period. Exceptions were LONG COVID symptoms (Endpoint #17) and significant cardiovascular events (Endpoints #20 & 22), both monitored until Week 24.
Description: To avoid duplicating data between the AE log and the LONG COVID symptom log, all the LONG COVID symptoms (core and non-core) were only entered in the LONG COVID symptom log even if they appeared or worsened after the baseline inventory. However, if a LONG COVID symptom appeared or worsened after the baseline inventory and is unexpected and/or exceeded in severity the normal LONG COVID evolution, then the said symptom were to be entered on the AE log during the AE collection period.
Arm/Group | LAU-7b for 3 Cycles (Arm 1, AAA) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) | Placebo for 3 Cycles (Arm 3, PPP)
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/91 | 0/90
Serious Adverse Events (participants affected / at risk) | 1/90 | 2/91 | 2/90
Other Adverse Events (participants affected / at risk) | 71/90 | 71/91 | 59/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAU-7b for 3 Cycles (Arm 1, AAA) (N=90) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) (N=91) | Placebo for 3 Cycles (Arm 3, PPP) (N=90)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAU-7b for 3 Cycles (Arm 1, AAA) (N=90) | LAU-7b for 1 Cycle, Then Placebo (Arm 2, APP) (N=91) | Placebo for 3 Cycles (Arm 3, PPP) (N=90)
Dry eye (Eye disorders) | 11 (11) | 6 (8) | 2 (5)
Vision blurred (Eye disorders) | 2 (2) | 7 (10) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 6 (7) | 6 (6)
Constipation (Gastrointestinal disorders) | 10 (11) | 5 (5) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 17 (22) | 4 (4) | 9 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (10) | 7 (7) | 3 (4)
Nausea (Gastrointestinal disorders) | 7 (8) | 10 (13) | 8 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (8) | 3 (3)
Influenza like illness (General disorders) | 4 (4) | 3 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 8 (8) | 8 (8) | 9 (9)
Dizziness (Nervous system disorders) | 6 (6) | 8 (10) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 5 (7) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (14) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 5 (5) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT05999435/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT05999435/SAP_001.pdf